CLINICAL TRIAL: NCT04242615
Title: Acute Kidney Injury in Non-Critical Care Setting: Elaboration and Validation of an In-hospital Death Prognosis Score
Acronym: AKI-DPS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/455
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Intra-hospital Mortality; Epidemiological Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prognostic score cohort: 323 patients included between January 1, 2001 to December 31, 2004
  Interventions: Other: Prognostic score
- Prognostic score validation cohort: 534 patients included between January 1, 2010 to December 31, 2013
  Interventions: Other: Prognostic score

INTERVENTIONS:
Other: Prognostic score

SUMMARY:
Acute renal failure (AKI) is defined by a deterioration of kidney function over a short period. This definition was clarified recently in order to allow homogenization and optimal comparison of patients in clinical studies by the classifications RIFLE in 2004, AKIN in 2007 and KDIGO in 2013. These classifications decline several stages of ARI through the increase in the plasma creatinine level and the decrease in urine flow.

Even though AKI is a frequent pathology in all hospitalized patients, there are only few studies that are interested in this entity in conventional hospital services except intensive care or intensive care. Indeed, the recent meta-analysis including the 154 studies focusing on the ARI defined by the KDIGO criteria, only 7 have recruited patients in conventional nephrology services. However, patients admitted for an ARI which requires treatment in a medical service probably have epidemiological characteristics and a different prognosis than those requiring treatment in intensive care. In addition, the parameters of the RIFLE, AKIN or KDIGO scores are more difficult to establish in conventional hospital services than in intensive care, especially for hourly monitoring of urine flow, not allowing an optimal classification of the episode of IRA.

This study set out to develop a prognostic score for intra-hospital mortality in ARI based on a first historical cohort. The investigators then validated this score on a second prospective cohort obtained over an independent inclusion period and at a distance from the first.

ELIGIBILITY:
Inclusion Criteria:

* all patients over 18 years of age admitted for ARI, defined by an increase in serum creatinine of more than 50% of baseline serum creatinine in patients without chronic kidney disease or an increase in serum creatinine greater than 100 umol / L compared to baseline serum creatinine if the patient had a serum creatinine clearance less than 60 mL / min / 1.73m2 calculated by the MDRD formula (Modification of the Diet in Renal Disease), hospitalized in the Nephrology department of the Besançon University Hospital Center

Exclusion Criteria:

* kidney transplant and patients from an intensive care unit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: We included all patients over 18 years of age admitted for ARI, defined by an increase in serum creatinine of more than 50% of baseline serum creatinine in patients without chronic kidney disease or increased serum creatinine at 100 umol / L compared to baseline serum creatinine if the patient had a serum creatinine clearance less than 60 mL / min / 1.73m2 calculated by the MDRD (Modification of the Diet in Renal Disease) formula, hospitalized in the Nephrology department of the Besançon University Hospital Center. Our exclusion criteria were kidney transplantation and patients from the intensive care unit.
  In our analysis, we constituted two cohorts: the first from January 1, 2001 to December 31, 2004 for the development of the prognostic score, then a second extending from January 1 2010 to December 31, 2013 for the validation of the score.
Sampling Method: Non-Probability Sample
Enrollment: 857 (Actual)
Dates: Start 2001-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Risk of intra-hospital mortality | 4 years
  Association between the clinical and biological parameters collected at the entry of patients included in the first cohort and the risk of intra-hospital mortality

IPD SHARING:
Plan to Share IPD: Undecided